CLINICAL TRIAL: NCT02591602
Title: Teleradiology Program for Frail Patients Living at Home or in Nursing-homes
Acronym: RADHOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Vittoria Tibaldi, MD PhD, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: RF-2009 -1550148
Record Dates: First submitted 2015-09-25; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Telemedicine; Teleradiology; Cost-Benefit Analysis; Frail Elderly

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CASI (Experimental): Teleradiology service for patients residing at home or in nursing homes
  Interventions: Other: Teleradiology Service
- CONTROLLI (No Intervention): X-ray hospital department

INTERVENTIONS:
Other: Teleradiology Service — Teleradiology Service at home or in nursing homes
  Arms: CASI

SUMMARY:
Transporting radiology to the patient's home is challenging. Preliminary experiences conducted in Turin (Italy) and Lund (Sweden) indicate that the coupling of simple, light-weight X-ray equipments with a Computed radiography or Digital Radiography systems could be effective for externalization of radiographic service.

The image and examination quality has been proved to be the same than those performed with a stationary equipment and analysis on safety of radio-protection systems show a very low risk exposure for health staff as well as for the general population.

Mobile radiography in nursing homes has shown to be technically feasible and the most beneficial results were that patients avoided unnecessary transport back and forth to the hospital; in both experiences the majority of patients could be treated locally.

The key points of RADHOME project are two:

1. The first one is to built a network model, with the aim to disseminate clinical use of domiciliary radiology.
2. The second one is to demonstrate clinical efficiency and cost-effectiveness of domiciliary radiology.

DETAILED DESCRIPTION:
Europe currently has the highest proportion of older people in the world and is expected to maintain this leading position for the next 50 years.

Population ageing is a great challenge for public health care systems as well as for economic development. As nations age, the prevalence of disability, frailty, and chronic diseases is expected to increase dramatically.

The hospital, which at the moment is the first choice for the delivery of acute medical care, is not an ideal environment for frail, elderly patients. New functional impairment and iatrogenic events such as nosocomial infections, pressure sores, falls and delirium, are common during hospital stay.

With developments in medical and other technologies, people with very complex conditions can increasingly have the possibility to remain at home or in nursing homes rather than in hospital.

Technologies can also improve the quality of life of patients and informal caregivers, allowing people to receive care and remain active at home and in the community, instead of being institutionalized.

These societal changes, such as needs of health care cost reduction and an aging population, are the main driving force for the development of telemedicine, especially for elderly patients.

Residents in nursing homes or patients treated at home by community care services are usually old or very old, multimorbid and often cognitively impaired. For these patients transportation to the hospital for X-ray examinations may be an exhausting and disorienting experience. They are collected by an ambulance or taxi and taken away from their environment and people they know. Patients wait in hospital corridors to have a fairly simple X-ray done and then wait for the pickup.

The first objective of RADHOME is to move equipments instead of patients in order to give a response to the geriatric tsunami and to the demand for more flexible health services, providing a view to advancing the economic efficiency of this service.

Teleradiology has become an essential part of the practice of radiology, with broad implications for care delivery and the organization of work: combining teleradiology and domiciliary X-ray examination has the potential to greatly improve the quality of care for elderly frail patients with acute or chronic conditions.

Until now no wide randomized study on radiology at home has been published. Hence main aim of this project is to carefully analyze feasibility, safety and cost-effectiveness of a public, extra-hospital and domiciliary radiology service for frail elderly or immobile patients, more vulnerable to environmental and social changes than other groups of patients, which health conditions discourage the transportation to hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients residents in nursing homes
* patients cared at home by community care services
* immobilization or chairbound
* need for chest, pelvis/hips, joints, upper and lower limbs, hands and feet X-rays,

Exclusion Criteria:

* need of urgent examination (within24 hours)
* need of X-ray examinations not suitable at home/nursing home.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical impact of the activation of a teleradiology service for home care teams and nursing homes - number of participants with positive clinical impact as assessed by multidimensional assessment. | 4 years
  All patients will be examinated using a standardized protocol which included multidimensional assessment. The multidimensional evaluation will be performed using standardized instruments: Activities of Daily Living (ADL) and Instrumental Activity of Daily Living (IADL) for functional status, Geriatric Depression Scale (GDS) for depression, Mini Mental State Examination (MMSE) for cognitive status, Cumulative Illness Rating Scale (CIRS) for comorbidity, Confusion Assessment Method (CAM) for delirium. A pain evaluation will be performed using the Visual Analogic Scale (VNS).

SECONDARY OUTCOMES:
Organizational impact of the activation of a teleradiology service for home care teams and nursing homes - waiting time and organizational path. | 4 years
Economic impact of the activation of a teleradiology service for home care teams and nursing homes - cost effectiveness analysis. | 4 years
Number of participants with positive impact on life quality as assessed by Nottingham Health Profile (NHP) for quality of life. | 4 years
  Technology can also improve the quality of life of patients and informal carers, making it more likely that the people receiving care and their informal carers can continue to stay active at home and in the community instead of being institutionalized.
Number of patients and care givers with high degree of satisfaction as assessed by Parasuraman Servqual methods. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Vittoria Tibaldi, Medicine, Principal Investigator — A.O.U. Città della Salute e della Scienza